CLINICAL TRIAL: NCT00477828
Title: Cognitive Benefits of Treating Apnea in Dementia
Brief Title: Effect of Treating Sleep Apnea on Cognition in Patients With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01AG008415 (NIH)
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2007-05

CONDITIONS: Dementia; Sleep Apnea
Keywords: sleep apnea; dementia; excessive sleepiness; cognition
MeSH Terms: conditions — Dementia; Sleep Apnea Syndromes; Disorders of Excessive Somnolence | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Continuous positive airway pressure

SUMMARY:
The purpose of this study is to determine whether treating sleep apnea with continuous positive airway pressure would result in improvements in cognition in patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Patients with sleep disordered breathing (SDB) experience nighttime sleep fragmentation and often become hypoxic during the night. The fragmentation and hypoxemia can frequently result in daytime impairments including impairments in cognitive functioning. The state-of-the-art treatment for SDB is Continuous Positive Airway Pressure (CPAP). Many SDB patients who are successfully treated with CPAP show improvement in memory and other cognitive functions. Data have shown that there is a strong relationship between SDB and dementia with patients with Alzheimer's Disease (AD) having a high rate of SDB. This proposal will examine whether treating SDB with CPAP in patients with AD will result in improvement in cognitive functioning. The specific aims are to assess whether patients with mild AD and SDB will tolerate CPAP and be compliant with treatment; to examine the effect of CPAP treatment on SDB in patients with mild AD and SDB; to examine the effect of CPAP treatment on cognitive functioning in patients with mild AD and SDB; to examine whether improvement is greater after six weeks of CPAP treatment than after three weeks of treatment. Since caregivers are often disturbed by the patients poor sleep, we will also evaluate the effect of the patients' treatment on their caregivers. Specifically, the secondary aims are to evaluate whether caregivers feel that CPAP improves the patient's sleep and to evaluate whether caregivers feel that their own sleep improves as the patient's sleep improves. Patient identified as having mild AD and SDB will have an extensive neuropsychological battery. Half will be randomized to CPAP treatment and the other half to shamCPAP. After three weeks neuropsychological tests will be repeated. The shamCPAP will be switched to CPAP and the CPAP group will remain on CPAP for an additional three weeks. Neuropsychological tests will again be repeated. The long-term goal of this line of research is to find a new approach that might improve the quality of life, delay the dementing process, postpone institutionalization and save millions of dollars in nursing care costs.

ELIGIBILITY:
Inclusion Criteria:

* Mild probable Alzheimer's disease (diagnosed according to the National Institute of Neurological and Communicative Disorders & Stroke-Alzheimer's Disease and Related Disorders Association [NINCDS-ADRDA] criteria).
* Mini Mental Status Exam score between 20 and 27
* Respiratory disturbance index >15 (i.e., 15 apneas plus hypopneas per hour of sleep) - Between the ages of 50-85 years
* Stable health
* reliable caregiver
* English speaking
* Patients will be allowed to continue acetylcholinesterase inhibitors, psychotropic medications, memory enhancers, health food supplements, etc. as long as they have been stable on the same dose for at least two months prior to participation and agree to continue on this dose for the duration of the study.

Exclusion Criteria:

* Currently receiving treatment for sleep apnea.
* Apneas primarily central in origin; narcolepsy or other sleep disorders
* Medication known to influence sleep (i.e. sedative hypnotics, narcotics) will be excluded if the dose can not remain stable and unchanged for the duration of the study.
* Bronchospastic and symptomatic chronic obstructive pulmonary disease as indicated by regular use of bronchodilators, steroids, history of carbon dioxide retention, waking hypoxemia (PaO2 <60 mmHg or SpO2 <92 % by pulse oximetry), or use of supplemental oxygen.
* Symptomatic coronary or cerebral vascular disease (history of myocardial infarction, angina, stroke, or transient ischemic attacks), history of life-threatening arrhythmias, cardiomyopathy, history of psychosis, or current alcohol or drug abuse
* Current diagnosis of active uncontrolled seizure disorder
* Any other advanced, severe and unstable disease of any type that may put the subject at special risk or interfere with primary and secondary variable evaluations
* Change in any medication within one month of participation.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2000-04; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
cognitive functioning; reports of daytime sleepiness; reports of quality of sleep | three weeks

SECONDARY OUTCOMES:
Caregivers' reports about their sleep | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Ancoli-Israel, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Result] Cooke JR, Liu L, Natarajan L, He F, Marler M, Loredo JS, Corey-Bloom J, Palmer BW, Greenfield D, Ancoli-Israel S. The effect of sleep-disordered breathing on stages of sleep in patients with Alzheimer's disease. Behav Sleep Med. 2006;4(4):219-27. doi: 10.1207/s15402010bsm0404_2. PMID 17083302
- [Result] Cooke JR, Loredo JS, Liu L, Marler M, Corey-Bloom J, Fiorentino L, Harrison T, Ancoli-Israel S. Acetylcholinesterase inhibitors and sleep architecture in patients with Alzheimer's disease. Drugs Aging. 2006;23(6):503-11. doi: 10.2165/00002512-200623060-00005. PMID 16872233
- [Result] Chong MS, Ayalon L, Marler M, Loredo JS, Corey-Bloom J, Palmer BW, Liu L, Ancoli-Israel S. Continuous positive airway pressure reduces subjective daytime sleepiness in patients with mild to moderate Alzheimer's disease with sleep disordered breathing. J Am Geriatr Soc. 2006 May;54(5):777-81. doi: 10.1111/j.1532-5415.2006.00694.x. PMID 16696743
- [Result] Ayalon L, Ancoli-Israel S, Stepnowsky C, Marler M, Palmer BW, Liu L, Loredo JS, Corey-Bloom J, Greenfield D, Cooke J. Adherence to continuous positive airway pressure treatment in patients with Alzheimer's disease and obstructive sleep apnea. Am J Geriatr Psychiatry. 2006 Feb;14(2):176-80. doi: 10.1097/01.JGP.0000192484.12684.cd. PMID 16473983
- [Derived] Ancoli-Israel S, Palmer BW, Cooke JR, Corey-Bloom J, Fiorentino L, Natarajan L, Liu L, Ayalon L, He F, Loredo JS. Cognitive effects of treating obstructive sleep apnea in Alzheimer's disease: a randomized controlled study. J Am Geriatr Soc. 2008 Nov;56(11):2076-81. doi: 10.1111/j.1532-5415.2008.01934.x. Epub 2008 Sep 15. PMID 18795985